CLINICAL TRIAL: NCT07037238
Title: An Open-Label, Single-Arm Exploratory Clinical Study of Everolimus for the Treatment of Vascular Malformations
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hongtao1
Record Dates: First submitted 2025-05-27; First posted 2025-06-25 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Vascular Malformations
Keywords: Vascular malformations; mTOR Inhibitors; Pharmacological Treatment
MeSH Terms: conditions — Vascular Malformations | interventions — Everolimus

STUDY DESIGN:
Intervention Model Description: A total of 10 participants aged 18 to 65 years with a confirmed diagnosis of vascular malformation will be enrolled. Eligible patients must be deemed by the investigator to be unsuitable for effective surgical treatment. After screening, qualified participants will receive oral everolimus once daily in continuous cycles of 28 days. The daily dosage of everolimus for adult patients will be 10 mg. Treatment will continue until disease progression, intolerable toxicity, lack of clinical benefit as determined by the investigator, study termination, or any other pre-defined discontinuation criteria-whichever occurs first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- An Open-Label, Single-Arm Exploratory Study of Everolimus (Experimental): Subjects will receive everolimus 10 mg orally once daily in continuous 28-day treatment cycles, until the occurrence of disease progression, intolerable toxicity, lack of clinical benefit as determined by the investigator, end of study, or other protocol-specified criteria for treatment discontinuation (whichever occurs first).
  Interventions: Drug: Everolimus 10mg daily

INTERVENTIONS:
Drug: Everolimus 10mg daily — An oral mTOR inhibitor

SUMMARY:
This study is a single-arm exploratory trial conducted by Xuanwu Hospital, Capital Medical University, aiming to evaluate the efficacy and safety of everolimus monotherapy in adult patients with vascular malformations.

DETAILED DESCRIPTION:
This study is a single-arm exploratory trial designed to evaluate the efficacy and safety of everolimus monotherapy in adult patients with vascular malformations.

A total of 10 participants aged 18 to 65 years with a confirmed diagnosis of vascular malformation will be enrolled. Eligible patients must be deemed by the investigator to be unsuitable for effective surgical treatment. After screening, qualified participants will receive oral everolimus once daily in continuous cycles of 28 days. The daily dosage of everolimus for adult patients will be 10 mg. Treatment will continue until disease progression, intolerable toxicity, lack of clinical benefit as determined by the investigator, study termination, or any other pre-defined discontinuation criteria-whichever occurs first.

The primary objective of this study is to assess the therapeutic efficacy of everolimus in patients with vascular malformations, primarily through evaluation of lesion volume using MRI sequences. All participants will undergo MRI-based target lesion volume analysis and assessments of microbleeding, iron deposition, and hemorrhage risk during the screening period, at the end of treatment cycles 3, 6, and 12, every 6 cycles thereafter, and at the end-of-treatment (EOT) visit. Clinical signs, symptom scores, and quality-of-life improvements will also be evaluated. The acceptable window for these assessments is ±7 days. If a participant has not undergone efficacy evaluation within 3 months, a final assessment should be conducted at the EOT visit.

ELIGIBILITY:
Inclusion Criteria

* Patients aged ≥18 and ≤65 years;
* No gender restrictions;
* Diagnosed with vascular malformation by MRI;
* No major surgery within the past 3 months;
* Able to swallow and retain oral medication, with no significant gastrointestinal abnormalities that may affect drug absorption, such as malabsorption syndrome, intestinal obstruction, or extensive gastrointestinal resection;
* Able to provide peripheral blood samples for biomarker testing at a central laboratory;
* Patients must have adequate organ and bone marrow function, and must not have received blood transfusions or any supportive treatments (e.g., cytokines or erythropoietin) to increase white blood cells, platelets, or hemoglobin levels within 7 days before screening tests:Absolute neutrophil count ≥1.0×10⁹/L;Hemoglobin ≥90 g/L; Platelets ≥100×10⁹/L;Total bilirubin ≤1.5× upper limit of normal (ULN), or ≤3.0× ULN for patients with Gilbert's syndrome;AST and ALT ≤2.5× ULN;Albumin ≥3 g/dL; Serum creatinine <1.5× ULN or creatinine clearance ≥50 mL/min;Urine protein <2+; if ≥2+, then 24-hour urine protein must be ≤1 g;Coagulation: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤1.5× ULN.
* Patients must voluntarily sign the written informed consent form and be able to complete follow-up;
* For patients of childbearing potential: they must agree to use highly effective contraceptive methods, such as combined hormonal contraception, progestogen-only hormonal contraception associated with ovulation inhibition, intrauterine devices (IUDs), intrauterine hormonal systems (IUS), bilateral tubal occlusion, or partner vasectomy, or to practice sexual abstinence during the treatment period and for at least 90 days after the last dose. Male patients must agree to refrain from sperm donation for at least 90 days after the last dose.

Exclusion Criteria:

* Diagnosed with Hereditary Hemorrhagic Telangiectasia (HHT), Arteriovenous Malformation (AVM), or PTEN Hamartoma Tumor Syndrome (PHTS);
* Patients who have previously received any of the following treatments after birth: participation in other interventional clinical trials targeting cerebral cavernous malformations (CM);
* Presence of malignant tumors currently or within the past three years, except for curatively treated non-melanoma skin basal cell carcinoma, ductal carcinoma in situ of the breast, or cervical carcinoma in situ;
* Unable to undergo MRI scans and/or have contraindications for MRI (e.g., interference from prosthetics, orthodontic devices, etc., affecting target lesion volume analysis on MRI);
* Modified Rankin Scale (mRS) score of 5, respiratory failure, or currently experiencing severe bleeding requiring life-support treatment;
* Severe renal failure (e.g., creatinine clearance \[CrCl] < 30 mL/min, or significantly elevated serum creatinine not correctable by other means), recent history (within past 3 months) of renal failure or end-stage renal disease without effective treatment, or currently undergoing dialysis;
* Severe hepatic failure, including but not limited to: Child-Pugh Class C or higher, recent (within 3 months) uncontrolled symptoms related to hepatic failure such as ascites, jaundice, coagulopathy, or hepatic encephalopathy, or patients requiring liver transplantation;
* Currently using other immunosuppressants or patients with immunodeficiency;
* Patients requiring use of medications that interfere with or inhibit CYP3A4 enzyme activity, or medications such as cisapride or metoclopramide;
* Patients with dysphagia, active gastrointestinal disorders, malabsorption syndrome, or other conditions that may affect the absorption of the investigational drug;
* Interstitial pneumonitis, including clinically significant radiation pneumonitis;
* Severe asthma;
* Uncontrolled diabetes mellitus;
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements;
* First-degree relatives with a history of sudden cardiac death before the age of 50. First-degree relatives are defined as those with a direct bloodline, such as parents and children, grandparents and grandchildren, or maternal grandparents and maternal grandchildren;
* Active bacterial, fungal, or viral infections, including active hepatitis B (HBsAg positive with HBV DNA > 1000 IU/mL or meeting local diagnostic criteria for active HBV infection), hepatitis C (HCV RNA positive), or HIV infection (HIV positive);
* Pregnant or breastfeeding women. Any patient who becomes pregnant during the trial must withdraw from the study;
* Known hypersensitivity to everolimus, other rapamycin derivatives, or any of the excipients in this product. Observed allergic reactions to everolimus or related compounds include but are not limited to: hypersensitivity, dyspnea, flushing, chest pain, or angioedema (e.g., airway or tongue swelling with or without respiratory compromise);
* Other factors, as determined by the investigator, that may lead to early study termination, such as presence of other severe diseases (including psychiatric disorders) requiring concomitant treatment, significantly abnormal lab values, or social/family issues that may affect patient safety or data collection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) assessed by MRI | 1 year

SECONDARY OUTCOMES:
Duration of Response (DOR) and 1-year DOR rate assessed by MRI | 1 year
Mean Percentage Reduction in Target Lesion Volume at 3, 6, and 12 Months Assessed by MRI | 1 year
Changes in Perilesional Microbleeds and Iron Deposition at 3, 6, and 12 Months Assessed by MRI QSM Sequence. | 1 year
Changes in lesion hemorrhage risk during the follow-up period | 1 year
  Based on MRI, imaging evidence of hemorrhage was defined as changes meeting the following criteria: (1) an increase in lesion size or alteration in its shape; and (2) a change in signal intensity, primarily characterized by a shift from hypointensity to hyperintensity, especially on T1-weighted sequences. Hemorrhage rates were calculated at 3, 6, and 12 months during follow-up to comprehensively evaluate the temporal changes in hemorrhagic risk of the lesion.
The frequency and severity of intracranial hemorrhage events during the follow-up period were assessed through clinical records, imaging examinations (MRI), and the mRS scoring system. | 1 year
Changes in patients' clinical signs and symptom scores from baseline. | 1 year
  The effectiveness of the medication and patient prognosis were comprehensively assessed by comparing the clinical symptoms and mRS scores of patients after treatment with baseline clinical symptoms and mRS scores. The mRS scale ranges from 0 to 5, with a decrease in score indicating a more favorable prognosis.
Disease Control Rate (DCR) assessed by MRI | 1 year
Progression-Free Survival (PFS) and 1-year PFS rate assessed by MRI | 1 year
The frequency and types of seizures during the follow-up period were recorded and assessed through seizure event logs and classification of seizure types. | 1 year

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 1year
  The type and frequency of treatment-emergent adverse events (TEAEs) occurring during the treatment period, evaluated according to NCI-CTCAE version 5.0;Treatment-related TEAEs;Serious adverse events (SAEs);TEAEs leading to permanent discontinuation of treatment;Incidence and frequency of death occurring within 30 days after the last dose of treatment;Laboratory abnormalities assessed according to NCI-CTCAE version 5.0.
Changes in patients' FACIT scores during the follow-up period | 1year
  The change in the patient's quality of life compared to baseline was primarily assessed using the Functional Assessment of Chronic Illness Therapy (FACIT) system. The score ranges from 0 to 108, and the scale is divided into four parts: Physical Well-Being (PWB), Social and Family Well-Being (SWB), Emotional Well-Being (EWB), and Functional Well-Being (FWB). Among these, lower scores in Physical Well-Being and Emotional Well-Being indicate better quality of life and prognosis, while higher scores in Social and Family Well-Being and Functional Well-Being indicate better quality of life and prognosis.
Pharmacokinetic (PK) profile/parameters | 1 year
  In this study, we will evaluate the pharmacokinetic (PK) profile of the drug by measuring "peak plasma concentration (Cmax)" over the one-year treatment period to assess the drug's metabolic behavior.
Pharmacokinetic (PK) profile/parameters | 1 year
  In this study, we will assess the pharmacokinetic (PK) profile of the drug by measuring the area under the plasma concentration versus time curve (AUC) over the one-year treatment period to evaluate the drug's metabolic characteristics.
Changes in patients' mRS scores during the follow-up period | 1year
  The change in the patient's quality of life compared to baseline was primarily assessed using the Modified Rankin Scale (mRS) score. The mRS score ranges from 0 to 5, with lower scores indicating better functional status, higher quality of life, and a better prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- the Department of Neurosurgery, China International Neuroscience Institute, Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
From 6 months post analysis and article publication, the following will be made available long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept Department of Neurosurgery, Xuanwu Hospital, Capital Medical University conditions for access:
  * Individual participant data that underlie the results reported in this article after de- identification
  * Trial protocol,Statistical Analysis Plan,PICF The Sponsor-Investigator will be the long-term custodian after the archive period has finished.
Supporting Information: Study Protocol
Time Frame: Available from 6 months following analysis and article publication
Access Criteria: Future researchers must be from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept Department of Neurosurgery, Xuanwu Hospital, Capital Medical University's conditions for access
URL: https://www.xwhosp.com.cn/